CLINICAL TRIAL: NCT00418509
Title: A Randomized, Single Dose, 3-Period Crossover Study to Evaluate the Dosage Form Proportionality, Dose Proportionality and Pharmacokinetics of Mometasone Furoate and Formoterol Fumarate From Three Combination MDI Formulations
Brief Title: Study of Mometasone Furoate/Formoterol Fumarate Inhalation Combination in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CFOR258H2104
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Dose proportionality; pharmacokinetics; mometasone; formoterol; Healthy volunteers study
MeSH Terms: interventions — Mometasone Furoate; Formoterol Fumarate

INTERVENTIONS:
Drug: Mometasone furoate
Drug: Formoterol fumarate

SUMMARY:
This study will compare the performance of three combination metered dose inhalation devices and the variability of mometasone and formoterol doses delivered to the lungs in a healthy volunteer population

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects age 18 to 65 years of age (included)
* In good health as confirmed by past medical history
* Female subjects must be either surgically sterilized at least 6 months prior to study participation or post-menopausal (no regular menstrual bleeding for at least 2 years)
* Body mass index (BMI) within the range of 18.5 to 32 kg/m2 and weigh at least 50 kg
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Understand and sign the written informed consent

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 1 year with a pack year history of no greater than 10 pack years).
* Female subjects who are pregnant, or lactating
* Treatment with any oral or intravenous corticosteroids within 1 month of the first study treatment.
* Patients with a current respiratory tract infection or one within 1 month prior to screening.
* Patients with a history of malignancy, myocardial infarction, untoward reactions to sympathomimetic amines or inhaled medicine.

Subjects with a current or history of a clinically significant cardiac arrhythmia.

* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* A past medical history of clinically significant ECG abnormalities.
* History of fainting, known hypersensitivity to the study drug or drugs similar to the study drug. any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study, immunocompromise, including a positive HIV (ELISA and Western blot) test result, positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result, drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening evaluations.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-11

PRIMARY OUTCOMES:
Dosage form and dose proportionality of mometasone and formoterol from combination metered dose inhalers (MDI).

SECONDARY OUTCOMES:
Extrapulmonary (systemic) effects and safety of mometasone and formoterol from combination MDI formulations.
Plasma and urine concentrations mometasone and formoterol

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis, Horsham, United Kingdom